CLINICAL TRIAL: NCT07190222
Title: A Phase 2b/3, Randomized, Double-blind, Placebo-controlled, Multicenter Study, to Investigate the Efficacy and Safety of Lunsekimig in Adult Participants With Inadequately Controlled Chronic Obstructive Pulmonary Disease (COPD) Characterized by an Eosinophilic Phenotype
Brief Title: Efficacy, Safety, and Tolerability Study of Lunsekimig Compared With Placebo in Adult Participants With Inadequately Controlled Chronic Obstructive Pulmonary Disease (COPD), Characterized by an Eosinophilic Phenotype
Acronym: THESEUS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC18244; 2024-518213-25-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lunsekimig dose regimen A (Experimental): Participants will receive lunsekimig dose regimen A.
  Interventions: Drug: Lunsekimig
- Lunsekimig dose regimen B (Experimental): Participants will receive lunsekimig dose regimen B.
  Interventions: Drug: Lunsekimig
- Placebo (Placebo Comparator): Participants will receive lunsekimig-matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lunsekimig — Pharmaceutical form: solution for injection in prefilled syringe - Route of administration: Subcutaneous injection
  Other Names: SAR443765
  Arms: Lunsekimig dose regimen A; Lunsekimig dose regimen B
Drug: Placebo — Pharmaceutical form:s olution for injection - Route of administration: Subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a parallel, Phase 2/Phase 3, 3-arm study to investigate the efficacy, safety, and tolerability of subcutaneous (SC) treatment with lunsekimig compared with placebo in adult participants (aged 40 to 80 years, inclusive) with inadequately controlled Chronic obstructive pulmonary disease (COPD) characterized by an eosinophilic phenotype.

Participation to the study consists of 3 periods:

* Screening period of up to 4 weeks
* Randomized intervention period of approximately 48 weeks
* Follow-up period: Approximately 8 weeks The study duration will be up to 60 weeks.

DETAILED DESCRIPTION:
All eligible participants will undergo subcutaneous administrations of lunsekimig or matching placebo during a 48-weeks treatment period

ELIGIBILITY:
Inclusion Criteria:

* Between 40 to 80 years of age
* Physician diagnosed chronic obstructive pulmonary disease (COPD) ≥1 year
* Post-bronchodilator forced expiratory volume in 1 second (post-BD FEV1) ≥ 20% and ≤ 70% of predicted value and FEV1/FVC (forced expiratory volume in 1 second /forced vital capacity) <0.70
* Former or current smokers ≥10 pack-years
* Chronic Airways Assessment Test (CAAT) ≥10
* ≥2 moderate or ≥1 severe COPD exacerbations in the prior year
* Triple (ICS+LABA+LAMA) COPD therapy ≥12 consecutive weeks
* EOS (blood eosinophil count) ≥ 150 cells/μL
* 18.0 ≤ Body Mass Index ≤ 40.0 kg/m2

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Asthma, including pediatric asthma, or ACOS
* Significant pulmonary disease other than COPD
* Long-term oxygen therapy >4.0 L/min or requirement of >2.0 L/minO2 saturation to maintain oxygen saturation >88%
* Unstable disorder that can impact participants safety or study outcomes
* Active or incompletely treated tuberculosis
* Current or past malignancies
* Concomitant therapies:

  * long-term macrolides or iPDE-4 unless on stable therapy for > 6 months
  * any biologic therapy or systemic immunosuppressant within 8 weeks or 5 half-lives prior to Screening

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 942 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2029-11-27 (Estimated); Study Completion 2030-01-22 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of moderatetosevere chronic obstructive pulmonary disease (COPD) exacerbations | From Baseline up to 48 weeks
  The annualized moderate or severe COPD exacerbation rate up to 48 weeks treatment period compared to placebo

SECONDARY OUTCOMES:
Change from baseline in post-Bronchodilator Forced Expiratory Volume in 1 second (post-BD FEV1) | From Baseline up to 48 weeks
  The post-Bronchodilator Forced Expiratory Volume in 1 second is defined as the volume of air exhaled from the lungs in the first second of a forced expiration
Change from baseline in pre-Bronchodilator Forced Expiratory Volume in 1 second (pre-BD FEV1) | From Baseline up to 48 weeks
  The pre-Bronchodilator Forced Expiratory Volume in 1 second is defined as the volume of air exhaled from the lungs in the first second of a forced expiration.
Change from baseline in the SGRQ-C total score | From Baseline up to 48 weeks
  The St. George's Respiratory Questionnaire for patients with chronic obstructive pulmonary disease is derived from the St. George's Respiratory Questionnaire (SGRQ) and is designed to measure and quantify health status in adult patients with chronic airflow limitation. A global score ranges from 0 to 100 with lower scores indicating better quality-of-life.
SGRQ responder defined as an improvement of ≥4 points in the SGRQ-C total score | From Baseline up to 48 weeks
Change from baseline in the Chronic airways assessment Test (CAAT) score | From Baseline up to 48 weeks
  The CAAT is an 8-item patient-reported outcome (PRO) measure designed to assess the impact of chronic airways diseases, including COPD, on patients' health status. The CAAT has a scoring range of 0-40, with higher scores indicating a greater impact of the disease on health status.
CAAT responder defined as an improvement of ≥2 points in the CAAT) total score | From Baseline up to 48 weeks
Change from baseline in the E-RS:COPD total score | From Baseline up to 48 weeks
  The Evaluating Respiratory Symptoms in Chronic Obstructive Pulmonary Disease (E-RS:COPD) is an 11-item patient-reported outcome (PRO) measure that evaluates the severity of respiratory symptoms in patients with stable COPD. The total score ranges from 0 to 40, with higher scores indicating more severe respiratory symptoms.
E-RS:COPD responder defined as an improvement of ≥2 points in the ERS:COPD total score | From Baseline up to 48 weeks
Annualized rate of severe COPD exacerbations | From Baseline up to 48 weeks
Time to first moderate or severe COPD exacerbation | From Baseline up to 48 weeks
  Time to first occurrence of moderate to severe COPD exacerbation up to 48 weeks
Time to first severe COPD exacerbation | From Baseline up to 48 weeks
  Time to first occurrence of severe COPD exacerbation up to 48 weeks
Incidence of participants with TEAEs, including AESIs, and SAEs | From Baseline up to 56
  Treatment-Emergent Adverse Events (TEAEs), Adverse events of Special Interest (AESIs), Serious Adverse Events (SAEs)
Incidence of potentially clinically significant laboratory abnormalities | From Baseline up to 56 weeks
Serum concentration of lunsekimig | From Baseline up to 56 weeks
Incidence and titer of antidrug antibodies (ADAs) | From Baseline up to 56 weeks

CONTACTS AND LOCATIONS:
Locations (117):
- United States (44):
  - Tucson Clinical Research Institute- Site Number : 8400006, Tucson, Arizona
  - Ark Clinical Research- Site Number : 8400113, Long Beach, California
  - California Medical Research Associates - Northridge- Site Number : 8400089, Northridge, California
  - Alpine Clinical Research Center - Boulder - 47th Street- Site Number : 8400005, Boulder, Colorado
  - Critical Care Pulmonary & Sleep Associates- Site Number : 8400081, Lakewood, Colorado
  - Finlay Medical Research - Greenacres- Site Number : 8400107, Greenacres City, Florida
  - Direct Helpers Research Center- Site Number : 8400057, Hialeah, Florida
  - Pulmonary Specialists of the Palm Beaches- Site Number : 8400017, Loxahatchee Groves, Florida
  - DL Research Solutions- Site Number : 8400140, Miami, Florida
  - Phoenix Medical Research - Miami - 24th Street- Site Number : 8400027, Miami, Florida
  - Professional Research Center- Site Number : 8400046, Miami, Florida
  - Research Institute of South Florida- Site Number : 8400028, Miami, Florida
  - Innovations Biotech- Site Number : 8400019, Miami, Florida
  - Florida Institute for Clinical Research- Site Number : 8400001, Orlando, Florida
  - Avanza Medical Research Center- Site Number : 8400015, Pensacola, Florida
  - Hull and Hull Medical Specialists- Site Number : 8400002, Plantation, Florida
  - Appalachian Clinical Research- Site Number : 8400060, Adairsville, Georgia
  - Christie Clinic in Champaign on University- Site Number : 8400023, Champaign, Illinois
  - Asha Clinical Research - Munster- Site Number : 8400115, Hammond, Indiana
  - Care Access - Shreveport - Youree Drive- Site Number : 8400007, Shreveport, Louisiana
  - Lucida Clinical Trials- Site Number : 8400101, New Bedford, Massachusetts
  - Vitalis Clinical Research Center- Site Number : 8400040, Allen Park, Michigan
  - Bolt Clinical Research- Site Number : 8400086, Brighton, Michigan
  - Hannibal Regional Healthcare System- Site Number : 8400035, Hannibal, Missouri
  - Excel Clinical Research - Las Vegas- Site Number : 8400070, Las Vegas, Nevada
  - AB Clinical Trials- Site Number : 8400075, Las Vegas, Nevada
  - Bioluminux Clinical Research New Jersey- Site Number : 8400037, Trenton, New Jersey
  - Mid Hudson Medical Research - New Windsor- Site Number : 8400004, New Windsor, New York
  - Piedmont Healthcare - Family Medicine- Site Number : 8400022, Statesville, North Carolina
  - All-Trials Clinical Research- Site Number : 8400008, Winston-Salem, North Carolina
  - Asthma & Allergy Center - Toledo- Site Number : 8400110, Toledo, Ohio
  - Layrek Clinical Research- Site Number : 8400066, Tulsa, Oklahoma
  - The Oregon Clinic, PC- Site Number : 8400065, Portland, Oregon
  - MedTrial- Site Number : 8400010, Columbia, South Carolina
  - Chattanooga Research and Medicine- Site Number : 8400026, Chattanooga, Tennessee
  - IntraCare- Site Number : 8400034, Dallas, Texas
  - Premier Pulmonary Critical Care and Sleep- Site Number : 8400111, Denison, Texas
  - El Paso Pulmonary Association- Site Number : 8400033, El Paso, Texas
  - Axsendo Clinical Research - Houston- Site Number : 8400054, Houston, Texas
  - SE Houston- Site Number : 8400120, Houston, Texas
  - Synergy Group US - Missouri City- Site Number : 8400119, Missouri City, Texas
  - Synergy Group US - Missouri City- Site Number : 8400133, Missouri City, Texas
  - Medrasa Clinical Research - Wylie- Site Number : 8400124, Wylie, Texas
  - Rheumatology & Pulmonary Clinic- Site Number : 8400012, Beckley, West Virginia
- Argentina (12):
  - Investigational Site Number : 0320011, Berazategui, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320005, Buenos Aires
  - Investigational Site Number : 0320006, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320012, Buenos Aires
  - Investigational Site Number : 0320003, Buenos Aires
  - Investigational Site Number : 0320009, Córdoba
  - Investigational Site Number : 0320007, Mendoza
  - Investigational Site Number : 0320008, Mendoza
  - Investigational Site Number : 0320010, Santa Fe
- Australia (3):
  - Investigational Site Number : 0360006, South Brisbane, Queensland
  - Investigational Site Number : 0360002, Traralgon, Victoria
  - Investigational Site Number : 0360001, Osborne Park, Western Australia
- Centro Multidisciplinar de Estudos Clínicos- Site Number : 0760001, São Bernardo do Campo, São Paulo, Brazil
- Canada (9):
  - Investigational Site Number : 1240051, Kelowna, British Columbia
  - Investigational Site Number : 1240052, North Vancouver, British Columbia
  - Investigational Site Number : 1240041, Windsor, Ontario
  - Investigational Site Number : 1240053, Québec, Quebec
  - Investigational Site Number : 1240050, Saint-Charles-Borromée, Quebec
  - Investigational Site Number : 1240054, Saint-Charles-Borromée, Quebec
  - Investigational Site Number : 1240049, Saint-Laurent, Quebec
  - Investigational Site Number : 1240048, Trois-Rivières, Quebec
  - Investigational Site Number : 1240042, Victoriaville, Quebec
- Chile (6):
  - Investigational Site Number : 1520006, Temuco, La Araucanía
  - Investigational Site Number : 1520004, Recoleta, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Viña del Mar, Región de Valparaíso
  - Investigational Site Number : 1520007, Chillán
- China (23):
  - Investigational Site Number : 1560079, Jingzhou, New South Wales
  - Investigational Site Number : 1560001, Beijing
  - Investigational Site Number : 1560090, Changde
  - Investigational Site Number : 1560052, Chengdu
  - Investigational Site Number : 1560074, Chongqing
  - Investigational Site Number : 1560051, Foshan
  - Investigational Site Number : 1560042, Ganzhou
  - Investigational Site Number : 1560015, Guangzhou
  - Investigational Site Number : 1560009, Hangzhou
  - Investigational Site Number : 1560021, Huzhou
  - Investigational Site Number : 1560055, Jinan
  - Investigational Site Number : 1560028, Jinan
  - Investigational Site Number : 1560077, Luoyang
  - Investigational Site Number : 1560018, Nanyang
  - Investigational Site Number : 1560073, Panjin
  - Investigational Site Number : 1560045, Quzhou
  - Investigational Site Number : 1560050, Shanghai
  - Investigational Site Number : 1560017, Shanghai
  - Investigational Site Number : 1560036, Wenzhou
  - Investigational Site Number : 1560071, Wuhan
  - Investigational Site Number : 1560006, Xinxiang
  - Investigational Site Number : 1560076, Yiyang
  - Investigational Site Number : 1560084, Zigong
- New Zealand (3):
  - Investigational Site Number : 5540003, Christchurch, Canterbury
  - Investigational Site Number : 5540002, Ebdentown, Wellington Region
  - Investigational Site Number : 5540001, Auckland
- South Korea (7):
  - Investigational Site Number : 4100007, Anyang-si, Gyeonggi-do
  - Investigational Site Number : 4100005, Daegu, Gyeongsangbuk-do
  - Investigational Site Number : 4100003, Jeonju, Jeollabuk-do
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100006, Seoul, Seoul-teukbyeolsi
- Investigational Site Number : 1580001, Kaohsiung City, Taiwan
- United Kingdom (8):
  - Investigational Site Number : 8260035, Milton Keynes, Buckinghamshire
  - Investigational Site Number : 8260007, London, England
  - Investigational Site Number : 8260006, Southampton, Hampshire
  - Investigational Site Number : 8260030, Salford, Manchester
  - Investigational Site Number : 8260013, Chertsey, Surrey
  - Investigational Site Number : 8260016, London
  - Investigational Site Number : 8260005, Reading
  - Investigational Site Number : 8260017, Rotherham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC18244 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26889&tenant=MT_SNY_9011